CLINICAL TRIAL: NCT00387530
Title: A Phase II Study of Phenylbutyrate and Valganciclovir in Epstein-Barr Virus Positive Tumors
Brief Title: Phenylbutyrate and Valganciclovir in Treating Patients With Relapsed or Refractory Epstein-Barr Virus-Positive Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD-050126; CDR0000504022 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-VAL-108
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer; Head and Neck Cancer; Lymphoma; Lymphoproliferative Disorder
Keywords: recurrent lymphoepithelioma of the nasopharynx; post-transplant lymphoproliferative disorder; adult nasal type extranodal NK/T-cell lymphoma; recurrent adult Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Head and Neck Neoplasms; Lymphoma; Lymphoproliferative Disorders; Lymphoma, Extranodal NK-T-Cell; Hodgkin Disease | interventions — 4-phenylbutyric acid; Valganciclovir; Polymerase Chain Reaction; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study of Biopsy (Other)
  Interventions: Drug: oral sodium phenylbutyrate; Drug: valganciclovir; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Procedure: biopsy

INTERVENTIONS:
Drug: oral sodium phenylbutyrate
Drug: valganciclovir
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Procedure: biopsy

SUMMARY:
RATIONALE: The Epstein-Barr virus can cause cancer and lymphoproliferative disorders. Valganciclovir is an antiviral drug that acts against the Epstein-Barr virus. Phenylbutyrate may make cells infected with Epstein-Barr virus more sensitive to valganciclovir. Giving phenylbutyrate together with valganciclovir may block the growth of Epstein-Barr virus-infected cells and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving phenylbutyrate together with valganciclovir works in treating patients with relapsed or refractory Epstein-Barr virus-positive cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of Epstein-Barr virus (EBV) lytic phase activation by BZLF1 expression in patients with relapsed or refractory, EBV-positive malignancies treated with phenylbutyrate.

Secondary

* Determine tumor responses in patients treated with phenylbutyrate followed by valganciclovir.
* Track serum EBV load by quantitative polymerase chain reaction and correlate changes with EBV lytic phase activation/tumor response.

OUTLINE: This is an open-label study.

Patients receive oral phenylbutyrate three times daily on days 1-21 and oral valganciclovir once or twice daily on days 4-21. Treatment repeats every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Patients undergo biopsy on day 3 of course 1. Serum Epstein-Barr virus DNA is analyzed for expression of BZLF1 and LMP2 by quantitative polymerase chain reaction on days 3 and 14 of course 1 and on day 1 of each subsequent course.

After completion of study treatment, patients are followed at 1 and 3 months.

PROJECTED ACCRUAL: A total of 14 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven Epstein-Barr virus (EBV)-positive malignancy

  * Must have tissue analysis to confirm EBV positivity

    * Archival tissue ≤ 1 year old may be used
* Any of the following malignancies:

  * WHO type II or III nasopharyngeal carcinoma
  * Post-transplant lymphoproliferative disorder
  * Nasal NK/T-cell lymphoma
  * Hodgkin's lymphoma
  * Lymphoepithelioma-variant gastric carcinoma
  * AIDS-related lymphomas

    * Patients with CNS non-Hodgkin's lymphoma must have tumor cells present in the cerebrospinal fluid (and assessable with lumbar puncture)
* Relapsed or refractory disease

  * Must have received and failed all prior potentially curative treatment for disease
  * Eligible only for salvage therapy
* Must have tumor tissue amenable for minimally invasive biopsy (e.g., fine-needle aspiration or bone marrow biopsy)

  * No brain tumors not amenable to biopsy
* CNS metastases allowed provided ≥ 2 weeks since prior radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute granulocyte count ≥ 500/mm³
* Platelet count ≥ 50,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 40 mL/min
* Recovered from uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Able to take medication orally or by gastrostomy tube
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 90 days after completion of study treatment
* No uncontrolled grade 1 symptomatic diarrhea (i.e., > 3 stools/day)
* No concurrent serious medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent cerebrospinal fluid drugs allowed
* No concurrent zidovudine for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Evidence of Epstein-Barr virus (EBV) lytic phase activation (expression of EBV antigens BZLF1 and LMP2) as assessed by biopsy on day 3 of course 1

SECONDARY OUTCOMES:
Tumor response in patients with measurable disease as assessed by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: William L. Read, MD, Study Chair — University of California, San Diego
Locations (1):
- Rebecca and John Moores UCSD Cancer Center, La Jolla, California, United States